CLINICAL TRIAL: NCT04948502
Title: A Multicenter, Randomized, Positive-controlled Clinical Trial to Verify the Efficacy and Safety of the SaExten Vena Cava Filter System in Prevention of Pulmonary Embolism
Brief Title: SaExten Vena Cava Filter System in Prevention of Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShenZhen KYD Biomedical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KYD SaExten Vena Cava Filter
Record Dates: First submitted 2021-06-23; First posted 2021-07-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; inferior vena cava filter; deep vein thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SaExten vena cava filter (Experimental): Manufacturer: ShenZhen KYD BioTech Co., Ltd., China. SaExten vena cava filter system is a retrievable filter system consisting of two parts: the vena cava filter and the delivering system. The vena cava filter is a mesh filtering device that prevents the formation of pulmonary embolism by filtering the thrombus. The SaExten vena cava filter can be inserted through jugular or femoral veins, and can be retrieved through jugular vein within 90 days or indwelled in vena cava permanently.
  Interventions: Device: SaExten vena cava filter system
- Denali inferior vena cava filter (Active Comparator): Manufacturer: C. R. BARD, Inc., USA
  Interventions: Device: Denali inferior vena cava filter

INTERVENTIONS:
Device: SaExten vena cava filter system — Subjects will undergo intervention, be implanted with a SaExten filter. The filter will be retrieved within 90 days or indwelled permanently, depending on the existence of thrombosis and the evaluation of the physician.
  Other Names: SaExten VCF system
  Arms: SaExten vena cava filter
Device: Denali inferior vena cava filter — Subjects will undergo intervention, be implanted with a Denali filter. The filter will be retrieved within 90 days or indwelled permanently, depending on the existence of thrombosis and the evaluation of the physician.
  Other Names: Denali IVCF
  Arms: Denali inferior vena cava filter

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SaExten vena cava filter (VCF) system (ShenZhen KYD BioTech Co., Ltd., China) in prevention of pulmonary embolism (PE).

This is a prospective, multicenter, randomized controlled, positive-controlled clinical trial, which will enroll 204 participants in total. Participants will undergo interventions with SaExten VCF System or Denali filter (C. R. BARD, Inc., USA).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of SaExten vena cava filter (VCF) system in prevention of pulmonary embolism (PE).

This is a prospective, multicenter, randomized controlled, positive-controlled clinical trial, which will enroll 204 participants in total, with 102 in each group. Participants will undergo interventions with SaExten VCF System or Denali filter, and be followed up to 12 months if the implantation is permanent, to evaluate the efficacy and safety of SaExten VCF System in prevention of PE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and life expectancy ≥ 12 months;
2. The diameter of inferior vena cava is between 18.0mm and 26.0mm;
3. Patients with acute (≤14 days of onset) proximal (inferior lumen, iliac, femoral, popliteal vein) deep vein thrombosis (DVT), or at risk of pulmonary embolism (PE) caused by thrombus detoxification, with or without symptoms of pulmonary embolism;
4. People at risk of pulmonary embolism (PE) meet at least one of the following conditions:

   * Patients with acute DVT who plan to undergo catheter-directed thrombolysis (CDT), percutaneous mechanical thrombectomy (PMT) or surgical thrombectomy;
   * Patients who have failed anticoagulant therapy, have recurrent PE and/or DVT, and have contraindications to anticoagulant therapy or are at serious risk of bleeding;
   * Floating thrombus in iliac, femoral vein or inferior vena cava;
   * Patients with high risk factors for acute DVT and PE who underwent abdominal, pelvic or lower limb surgery;
   * Patients with DVT who have already developed a large area of PE and are at risk of developing PE again;
   * DVT accompanied by serious heart and lung disease, pulmonary hypertension;
   * Severe injuries (such as hip fracture, etc.), accompanied by vascular endothelial injury, accompanied by blood hypercoagulability and anticoagulant therapy contraindications;
5. Those who can understand the purpose of the trial, cooperate with the follow-up, and sign the informed consent voluntarily.

Exclusion Criteria:

1. Patients with severe stenosis or deformity of the inferior vena cava or severe spinal deformity;
2. Patients with uncontrolled infectious diseases, purulent embolism or fat embolism;
3. Previous vena cava filter implantation history;
4. Thrombosis in the venous access required for the filter implantation;
5. Patients with severe liver and renal dysfunction (ALT>3 times the upper limit of normal; Creatinine>225umol/L);
6. Patients with known uncorrectable bleeding or severe coagulation disease;
7. Patients who are allergic to contrast agents, nickel and have contraindication to X-ray;
8. With disease causing difficulties in treatment and evaluation (such as septicemia, bacteremia, toxemia, severe metabolic disease, cancer metastasis, mental illness, etc.);
9. Malignant tumor patients;
10. Pregnant and lactating women, or those who is planning parenthood;
11. Participated in clinical trials of other drugs or medical devices before inclusion and haven't reach the end point time limit;
12. Persons considered by the investigator to be unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Clinical success rate of IVCF implantation | 6 months
  Clinical success requires the following three factors:
  * No clinical symptomatic pulmonary embolism occurred within 6 months after long-term filter implantation, which was confirmed by CT pulmonary angiography (CTPA); No clinical pulmonary embolism occurred between the time of filter implantation and the time of filter retrieval, which was confirmed by pulmonary angiography.
  * The IVCF was successfully implanted with satisfactory shape and position;
  * No filter fracture, no displacement over 20 mm , no inclination (> 15°) during implantation/retrieval, no IVC penetration, no thrombosis of the IVC, and no implant-related or operation-related deaths.

SECONDARY OUTCOMES:
Technical success rate of IVCF implantation | 1 day
  Successful filter implantation is defined as: The filter was successfully implanted with satisfactory shape and position, and no complications associated with the filter occurred during the operation procedure.
Clinical success rate of IVCF retrieval | 90 days
  Clinical success of filter recovery is defined as: The filter was successfully and completely removed from patients attempting to retrieve the filter within 90 days of filter implantation, without complications requiring clinical intervention.
Technical success rate of IVCF retrieval | 90 days
  Successful filter retrieval is defined as: the filter was successfully and completely removed in patients who attempted to retrieve the filter within 90 days after implantation, and no complications associated with the filter occured during the operation.
Evaluation of operation performance of filter and transporting system | 90 days
  Technical success of the filter and transporting system is defined as: during the operation, the marking and development of the transporting system were good, the filter was transported to the expected position of the vena cava smoothly, the preloaded filter was released completely, and all parts of the transporting system were removed from the body smoothly without falling off or breaking.
The combined incidence of filter displacement over 20 mm, fracture, tilt (> 15°) and IVC penetration within 6 months after implantation | 6 months
  These measures are used to describe the incidences of filter post-implantation.
Incidence of pulmonary embolism within 6 months after implantation. | 6 months
  It is used to describe the incidence of PE post-implantation.
The incidence of new or aggravated deep vein thrombosis within 6 months after implantation | 6 months
  It is used to describe the incidence of DVT post-implantation.
The incidence of compound clinical events of pulmonary embolism, IVC thrombosis, death, and recurrent deep venous thrombosis of lower limbs at 30 days, 3 months, and 6 months after vena cava filter implantation | 30 days, 3 months, and 6 months
  These measures are used to describe the incidence of PE, IVC thrombosis, death, and and recurrent DVT post-implantation.
The number of days from implantation to retrieval (for patients whose filters have been retrieved) | 90 days
  It is used to describe the time from IVC filter implantation to retrieval.

CONTACTS AND LOCATIONS:
Overall Officials: Guangqi Chang, Dr., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (16):
- China (16):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - Handan First Hospital, Handan, Hebei
  - Luoyang Orthopedic-Traumatological Hospital of Henan Province, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The People's Hospitai of Liaoning Province, Shenyang, Liaoning
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang